CLINICAL TRIAL: NCT02726620
Title: Decision Support for Intraoperative Low Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Jonathan Wanderer, Medical Director of Procedure Preparation Center, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 160131
Record Dates: First submitted 2016-03-28; First posted 2016-04-04 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-04

CONDITIONS: Hypotension
Keywords: Decision support; Decision Support Systems, Clinical; Decision Support Techniques; Hypotension; Intraoperative Hypotension; Acute Kidney Injury; Postoperative Mortality; Blood Pressure
MeSH Terms: conditions — Hypotension; Acute Kidney Injury | interventions — Anesthesia, General; Anesthesia, Conduction; Anesthesia, Spinal; Anesthesia, Epidural; Propofol; Sevoflurane; Desflurane; Isoflurane; Ephedrine; Phenylephrine; Norepinephrine; Epinephrine; Dobutamine; Dopamine; Isoproterenol; Milrinone; Atropine; Glycopyrrolate; Vasopressins; Terlipressin; Sodium Chloride; Ringer's Lactate; Plasma-lyte 148; Lidocaine; Bupivacaine; Levobupivacaine; Ropivacaine; Mepivacaine; Tetracaine; Prilocaine; Procaine; chloroprocaine; Benzocaine; Carticaine

STUDY DESIGN:
Intervention Model Description: It is an interrupted time-series of a decision support package intervention that aims to study the the effect of the decision support package on patient outcome. The effects of the individual decision support components of the package on healthcare provider behavior will be studied in a nested cluster-randomized trial: in the first month the attending anesthesiologists will be randomized to near-realtime notifications or feedback emails; in the second month in-room providers will be randomized to near-realtime notifications or feedback emails. Starting month four all providers will receive both near-realtime notifications and feedback emails.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypotension decision support (Experimental): The intervention period. Several decision support elements are implemented to notify anesthesia providers: attending anesthesiologists and in-room anesthesia providers of intraoperative hypotension (threshold of a mean arterial pressure below 60 mmHg). Two types of decision support will be implemented: near real-time decision support and feedback emails.
  Near real-time decision support elements will notify the anesthesia providers of a blood pressure drop below the threshold and display the associated increased risk of acute kidney injury. The notification is presented through the pager system for attending anesthesiologists and through the anesthesia information management system for the in-room anesthesia provider.
  All providers will be notified through email within 24 hours after the end of an anesthetic case, when the patient had an episode of intraoperative hypotension that is associated with an increased risk of organ injury due to organ ischemia.
  Interventions: Procedure: Attending real-time decision support; Procedure: In-room real-time decision support; Procedure: Attending feedback emails; Procedure: In-room provider feedback emails; Device: Anesthesia Information Management System (AIMS); Device: Perioperative Data Warehouse (PDW); Procedure: General anesthesia; Device: Pager system; Procedure: Central neuraxial anesthesia; Procedure: Non-cardiac surgery; Drug: Propofol; Drug: Sevoflurane; Drug: Desflurane; Drug: Isoflurane; Drug: Ephedrine; Drug: Phenylephrine; Drug: Norepinephrine; Drug: Epinephrine; Drug: Dobutamine; Drug: Dopamine; Drug: Isoproterenol; Drug: Milrinone; Drug: Atropine; Drug: Glycopyrrolate; Drug: Vasopressin; Drug: Terlipressin; Drug: Sodium Chloride 0.9%; Drug: Ringer's lactate; Drug: Hydroxyethyl starch solutions; Drug: Fresh Frozen Plasma; Drug: Packed Red Blood Cells; Drug: Albumin solutions; Drug: Plasma-Lyte; Drug: Lidocaine; Drug: Bupivacaine; Drug: Levobupivacaine; Drug: Ropivacaine; Drug: Mepivacaine; Drug: Tetracaine; Drug: Prilocaine; Drug: Procaine; Drug: Chloroprocaine; Drug: Benzocaine; Drug: Articaine
- Usual care group (Active Comparator): The 'before' period - or historic control group - during which no decision support for intraoperative hypotension was being used, also known as 'usual care'. This is the three year period prior to the intervention period (the 'Intraoperative hypotension decision support' arm).
  Interventions: Procedure: General anesthesia; Procedure: Central neuraxial anesthesia; Procedure: Non-cardiac surgery; Drug: Propofol; Drug: Sevoflurane; Drug: Desflurane; Drug: Isoflurane; Drug: Ephedrine; Drug: Phenylephrine; Drug: Norepinephrine; Drug: Epinephrine; Drug: Dobutamine; Drug: Dopamine; Drug: Isoproterenol; Drug: Milrinone; Drug: Atropine; Drug: Glycopyrrolate; Drug: Vasopressin; Drug: Terlipressin; Drug: Sodium Chloride 0.9%; Drug: Ringer's lactate; Drug: Hydroxyethyl starch solutions; Drug: Fresh Frozen Plasma; Drug: Packed Red Blood Cells; Drug: Albumin solutions; Drug: Plasma-Lyte; Drug: Lidocaine; Drug: Bupivacaine; Drug: Levobupivacaine; Drug: Ropivacaine; Drug: Mepivacaine; Drug: Tetracaine; Drug: Prilocaine; Drug: Procaine; Drug: Chloroprocaine; Drug: Benzocaine; Drug: Articaine

INTERVENTIONS:
Procedure: Attending real-time decision support — Near real-time decision support elements will notify the attending anesthesiologists of a blood pressure drop below the threshold for intraoperative hypotension (mean arterial pressure below 60 mmHg). The notification is presented through the pager system. The page will also display the associated increased risk of organ injury due to organ ischemia.
  Arms: Hypotension decision support
Procedure: In-room real-time decision support — Near real-time decision support elements will notify the in-room anesthesia provider of a blood pressure drop below the threshold for intraoperative hypotension (mean arterial pressure below 60 mmHg). The notification is presented through the anesthesia information management system. The decision support system will display the associated increased risk of organ injury due to organ ischemia.
  Arms: Hypotension decision support
Procedure: Attending feedback emails — Attending anesthesiologists will be notified through email within 24 hours after the end of an anesthetic case, when the patient had an episode of intraoperative hypotension (mean arterial pressure below 60 mmHg or lower for a particular duration) that is associated with an increased risk of organ injury due to organ ischemia.
  Arms: Hypotension decision support
Procedure: In-room provider feedback emails — In-room anesthesia providers will be notified through email within 24 hours after the end of an anesthetic case, when the patient had an episode of intraoperative hypotension (mean arterial pressure below 60 mmHg or lower for a particular duration) that is associated with an increased risk of organ injury due to organ ischemia.
  Arms: Hypotension decision support
Device: Anesthesia Information Management System (AIMS) — The anesthesia electronic record keeping system
  Arms: Hypotension decision support
Device: Perioperative Data Warehouse (PDW) — The data warehouse that is used to gather perioperative data and create user reports. In this instance the PDW will be used to send the postoperative feedback emails.
  Arms: Hypotension decision support
Procedure: General anesthesia — Any anesthetic drugs that are used to induce general anesthesia above the level of sedation.
Device: Pager system — The mobile pager system through which alerts can be sent
  Arms: Hypotension decision support
Procedure: Central neuraxial anesthesia — Regional anesthesia effectuated through the placement of local anesthetics around the nerves of the central nervous system, e.g. spinal anesthesia and epidural anesthesia.
  Other Names: Regional anesthesia; Spinal anesthesia; Intrathecal anesthesia; Subarachnoid anesthesia; Epidural anesthesia; Central neuraxial blockade
Procedure: Non-cardiac surgery — Any surgical intervention that is not aimed at surgical correction of the heart
Drug: Propofol — Anesthetic drug used to maintain general anesthesia
Drug: Sevoflurane — Anesthetic drug used to maintain general anesthesia
Drug: Desflurane — Anesthetic drug used to maintain general anesthesia
Drug: Isoflurane — Anesthetic drug used to maintain general anesthesia
Drug: Ephedrine — Cardiovascular drug used to treat intraoperative hypotension
Drug: Phenylephrine — Cardiovascular drug used to treat intraoperative hypotension
Drug: Norepinephrine — Cardiovascular drug used to treat intraoperative hypotension
Drug: Epinephrine — Cardiovascular drug used to treat intraoperative hypotension
Drug: Dobutamine — Cardiovascular drug used to treat intraoperative hypotension
Drug: Dopamine — Cardiovascular drug used to treat intraoperative hypotension
Drug: Isoproterenol — Cardiovascular drug used to treat intraoperative hypotension
Drug: Milrinone — Cardiovascular drug used to treat intraoperative hypotension
Drug: Atropine — Cardiovascular drugs used to treat intraoperative hypotension
Drug: Glycopyrrolate — Cardiovascular drug used to treat intraoperative hypotension
Drug: Vasopressin — Cardiovascular drug used to treat intraoperative hypotension
Drug: Terlipressin — Cardiovascular drug used to treat intraoperative hypotension
Drug: Sodium Chloride 0.9% — Intravenous fluid used to treat intraoperative hypotension
Drug: Ringer's lactate — Intravenous fluid used to treat intraoperative hypotension
Drug: Hydroxyethyl starch solutions — Intravenous fluid used to treat intraoperative hypotension
Drug: Fresh Frozen Plasma — Intravenous fluid used to treat intraoperative hypotension
Drug: Packed Red Blood Cells — Intravenous fluid used to treat intraoperative hypotension
Drug: Albumin solutions — Intravenous fluid used to treat intraoperative hypotension
Drug: Plasma-Lyte — Intravenous fluid used to treat intraoperative hypotension
Drug: Lidocaine — Local anesthetic used for central neuraxial anesthesia.
  Other Names: Lignocaine
Drug: Bupivacaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Levobupivacaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Ropivacaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Mepivacaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Tetracaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Prilocaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Procaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Chloroprocaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Benzocaine — Local anesthetic used for central neuraxial anesthesia.
Drug: Articaine — Local anesthetic used for central neuraxial anesthesia.

SUMMARY:
The purpose of this study is to determine whether a decision support system can improve the adherence to thresholds for low blood pressure by anesthesia providers, which in turn prevents their patients from having organ injury.

DETAILED DESCRIPTION:
Blood pressure management is an important part of anesthesia. Many factors contribute to a change in blood pressure during a surgical procedure, such as blood loss, manipulation by surgeons, and there are several mechanisms through which anesthesia itself changes blood pressure. Although a high blood pressure also occurs during anesthesia, most of these factors lower a patient's blood pressure. When a patient's blood pressure becomes too low, the internal organs become at risk of receiving not enough blood (low perfusion or hypoperfusion). This low perfusion state can result in organ damage (ischemia) because of an insufficient supply of oxygen and glucose. Hence the important task of anesthesia providers to maintain the blood pressure of patients, using a wide range of drugs and other interventions.

A big challenge in blood pressure management is to know when a low blood pressure indeed results in low perfusion of organs. There is a large variation between patients in how susceptible they are to low blood pressure, as well as a difference between the organs in how easily they are damaged because of low perfusion. Elder patients, or patients with preexisting hypertension, heart problems or other cardiovascular diseases are more prone to a low blood pressure and are more likely to develop organ ischemia when there is a low blood pressure. The kidneys, the heart and the brain are the organs that are most at risk of organ damage. As one cannot measure the perfusion states of individual organs in individual patients, it is very difficult to know 'how low to go' with a patient's blood pressure.

Recent studies have used large datasets of patients to demonstrate that there is statistical association between low blood pressure during surgery and various types of organ injury. As patients are already treated for low blood pressure by anesthesia providers, this suggests that patients have low organ perfusion states despite the current treatment standards. A patient's blood pressure is not simply a dial that can be adjusted to a specific level. Finding the right level of interventions can be difficult in some patients. Consequently, lower blood pressures are common in anesthesia, even with the current standards of blood pressure management.

In this proposed study the investigators will implement two forms of decision support to assist anesthesia providers in blood pressure management. The decision support aims to educate anesthesia providers about the risks of low blood pressures in direct relation to the patients that they treat. One form of decision support will provide automated notifications through pagers and through the anesthesia information management system. These automated notifications pop up when the patient's blood pressure drops below a level that is associated with a risk of organ injury, and thus alerts the anesthesia provider of the blood pressure and its associated risk. The second form of decision support will send a postoperative email the day after the procedure when the patient has had a low blood pressure for particular duration. This email then provides feedback to the anesthesia provider by informing them of the increased risks of organ injury that are associated with that low blood pressure.

The study will look at both a change in patient outcome and a change in blood pressure management and will be performed at the Vanderbilt University Medical Center (VUMC). The change in patient outcome will primarily be studied through the occurrence of acute kidney injury in the first days following the procedure at the VUMC. The change in blood pressure management (provider behavior) will be studied by observing the depth and duration of low pressures during anesthesia, and the number of interventions that have been used to treat the blood pressure. Patient outcome will be studied by comparison of a baseline phase - before the decision support is implemented and uses historic data- and the intervention phase - the period during which the intervention is active. Only routinely collected clinical data will be used for these analyses: no additional data collection is required.

As it is impossible to know which form of decision support will be the most effective, the first three months of the intervention period will be a 'nested cluster-randomized trial'. The anesthesia providers (not the patients) will be randomized to either the automated notifications or the feedback emails. After three months all anesthesia providers will receive both forms of decision support for the remainder of the intervention period. The reason why anesthesia providers are randomized only during the first three months is that cross-over or contamination between the two groups is expected. This contamination could make it impossible to study the effect of the decision support on patient outcome, as there will be no longer any difference between the study groups.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* Inpatients
* Scheduled for a non-cardiac surgical procedure under general or central neuraxial anesthesia

Exclusion Criteria:

* Pre-existing end-stage renal disease: operationalized as a preoperative need for dialysis
* The following surgical procedures: renal surgery, cardiac surgery, organ transplantation, ophthalmic surgery, endoscopic gastrointestinal procedures, and (interventional) radiologic procedures.
* small non-invasive or minimally-invasive procedures will also be excluded, operationalized as excluding procedures with a surgical time of less than twenty minutes.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22435 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Wanderer, MD, MPhil, Principal Investigator — Vanderbilt University Medical Center, Department of Anesthesiology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Historic Cohort - Three Years
Arm/Group | Usual Care Group | Hypotension Decision Support
Started | 17463 | 0
MAP < 65 mmHg: Primary Analysis (Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis.) | 15624 | 0
Completed | 17463 | 0
Not Completed | 0 | 0
Period: Month 1: Attending Randomization
Arm/Group | Usual Care Group | Hypotension Decision Support
Started | 0 | 485
MAP < 65 mmHg: Primary Analysis (Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis.) | 0 | 432
Correct IOH Notifications (The decision support notifications log matches the actual occurrens of intraoperative hypotension.) | 0 | 313
Completed | 0 | 485
Not Completed | 0 | 0
Period: Months 2-3: In-room Providers Randomized
Arm/Group | Usual Care Group | Hypotension Decision Support
Started | 0 | 1253
MAP < 65 mmHg: Primary Analysis (Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis.) | 0 | 1103
Correct IOH Notifications (The decision support notifications log matches the actual occurrens of intraoperative hypotension.) | 0 | 825
Completed | 0 | 1253
Not Completed | 0 | 0
Period: Through End of Study: All Interventions
Arm/Group | Usual Care Group | Hypotension Decision Support
Started | 0 | 3234
MAP < 65 mmHg: Primary Analysis (Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis.) | 0 | 2793
Correct IOH Notifications (The decision support notifications log matches the actual occurrens of intraoperative hypotension.) | 0 | 2072
Completed | 0 | 3234
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis based on the 'Completed' number of patients from the Participant Flow (including patients who did not have any mean arterial pressure < 65 mmHg). The 'Hypotension decision support' arm summarizes the last three periods from the Participant Flow section (the intervention periods).
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | Hypotension Decision Support | Total
Number analyzed (Participants) | 17463 | 4972 | 22435
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [64 to 74] | 68 [64 to 74] | 68 [64 to 74]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Incomplete patient demographics section resulted in a row population difference from the Overall.
  Participants
    number analyzed (Participants) | 17438 | 4963 | 22401
    Female | 7731 | 2141 | 9872
    Male | 9707 | 2822 | 12529
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 4 | 22
  Asian | 113 | 36 | 149
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1111 | 380 | 1491
  White | 15571 | 4348 | 19919
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 650 | 204 | 854
Region of Enrollment [Number; unit: participants]
  United States | 17463 | 4972 | 22435
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Body Mass Index (BMI) in kg/m^2 Population: Incorrect demographics data resulted in row population differences from overall.
  kg/m^2
    number analyzed (Participants) | 17306 | 4930 | 22236
    (all) | 28 [24 to 32] | 28 [24 to 32] | 28 [24 to 32]
ASA Class [Count of Participants; unit: Participants] — The ASA (American Society of Anesthesilogists) physical status classification system is a system for assessing the fitness of patients before surgery. This is assessed by the attending anesthesiologist and is recorded on the preprocedure anesthesia evaluation. ASA Class I corresponds to a healthy patient; ASA Class 2 corresponds to a patient with mild systemic disease; ASA Class 3 is a patient with severe systemic disease; ASA Class 4 a patient with severe systemic disease that is a constant threat to life; ASA Class 5 is a moribund patient who is not expected to survive without the operation.
  Participants
    ASA Class 1 | 74 | 16 | 90
    ASA Class 2 | 3109 | 765 | 3874
    ASA Class 3 | 12344 | 3578 | 15922
    ASA Class 4 | 1885 | 585 | 2470
    ASA Class 5 | 51 | 28 | 79
Hypertension [Count of Participants; unit: Participants] — Comorbidities present at baseline: essential hypertension Population: No preoperative data on comorbidities was available in a structured form, resulting in missings.
  Participants
    number analyzed (Participants) | 15718 | 4500 | 20218
    (all) | 11403 | 3348 | 14751
Cardiac disease [Count of Participants; unit: Participants] — Comorbidities present at baseline: cardiac disease (cardiac arrythmia, congestive heart failure, valvular heart disease) Population: No preoperative data on comorbidities was available in a structured form, resulting in missings.
  Participants
    number analyzed (Participants) | 15718 | 4500 | 20218
    (all) | 4843 | 1489 | 6332
Renal Disease [Count of Participants; unit: Participants] — Comorbidities present at baseline: renal disease (non-endstage renal failure) Population: No preoperative data on comorbidities was available in a structured form, resulting in missings.
  Participants
    number analyzed (Participants) | 15718 | 4500 | 20218
    (all) | 1432 | 511 | 1943
Peripheral vascular disease [Count of Participants; unit: Participants] — Comorbidities present at baseline: peripheral vascular disease Population: No preoperative data on comorbidities was available in a structured form, resulting in missings.
  Participants
    number analyzed (Participants) | 15718 | 4500 | 20218
    (all) | 1947 | 596 | 2543
Diabetes Mellitus [Count of Participants; unit: Participants] — Comorbidities present at baseline: diabetes mellitus (any type) Population: No preoperative data on comorbidities was available in a structured form, resulting in missings.
  Participants
    number analyzed (Participants) | 15718 | 4500 | 20218
    (all) | 4456 | 1296 | 5752
Type of anesthesia [Count of Participants; unit: Participants]
  General anesthesia | 17051 | 4750 | 21801
  Central neuraxial anesthesia | 412 | 222 | 634
Procedure urgency [Count of Participants; unit: Participants]
  Elective surgery | 16452 | 4631 | 21083
  Emergency surgery | 1011 | 341 | 1352
Procedure duration [Median (Inter-Quartile Range); unit: minutes] — Duration of the procedure in minutes.
  minutes | 201 [144 to 281] | 196 [143 to 271] | 200 [144 to 278]
Surgical service [Count of Participants; unit: Participants] — Surgical specialty of the primary surgeon
  Participants
    ENT | 1891 | 528 | 2419
    Gynecology | 113 | 30 | 143
    General surgery | 3638 | 1001 | 4639
    Neurosurgery | 2138 | 622 | 2760
    Orthopedic surgery | 4283 | 1222 | 5505
    Plastic surgery | 776 | 195 | 971
    Thoracic surgery | 1056 | 310 | 1366
    Urology | 2648 | 778 | 3426
    Vascular surgery | 920 | 286 | 1206
AKI risk based on IOH depth and duration [Count of Participants; unit: Participants] — Risk of Acute Kidney Injury based on the depth and duration of intraoperative hypotension as defined in the present study.
  Participants
    AKI risk: none | 3684 | 1174 | 4858
    AKI risk: mild | 6622 | 1985 | 8607
    AKI risk: moderate | 4290 | 1136 | 5426
    AKI risk: high | 2867 | 677 | 3544

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Acute Kidney Injury
Description: Postoperative Acute Kidney Injury (AKI), Stage I or higher according to the KDIGO criteria (Kidney Disease: Improving Global Outcomes). The staging will be based on serum creatinine values, as documentation of urine output is probably not sufficiently accurate. This will be the primary outcome for the Vanderbilt University Medical Center. The creatinine measurements are part of routine clinical care. Therefore, absence of creatinine postoperative measurements are considered to be 'no suspicion of kidney injury'. KDIGO defines AKI as any of the following: Increase in serum creatinine by 0.3mg/dL or more within 48 hours or Increase in serum creatinine to 1.5 times baseline or more within the last 7 days or Urine output less than 0.5 mL/kg/h for 6 hours. Stage 1 is 1.5-9x baseline or >0.3 increase; Stage 2 is 2-2.9x baseline; Stage 3 is 3x baseline, or increase to > 4, or initiation of renal replacement therapy.
Time Frame: Within 7 days after surgery
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section).
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants
  AKI stage I or greater | 1333 | 372
  No AKI - Confirmed by measurement | 9670 | 2785
  No postoperative creatinine measurement | 4621 | 1171

2. Secondary Outcome: 30-day Mortality
Description: Vanderbilt University Medical Center: combination of in-hospital mortality and 'alive-index' (which checks for visits to the hospital in the electronic healthcare record as indication of being alive at 30 days)
Time Frame: 30 days after surgery
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section). For a large group of patients no mortality information was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 4667 | 1285
Participants | 511 | 143

3. Secondary Outcome: In-hospital Mortality
Description: Hospital mortality rate during a single hospital admission after the surgery
Time Frame: All postoperative days during a single hospital admission, expected median of 5 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 487 | 137

4. Secondary Outcome: Postoperative Acute Kidney Injury Stage 2
Description: Postoperative Acute Kidney Injury (AKI), Stage II or higher according to the KDIGO criteria (Kidney Disease: Improving Global Outcomes). The staging will be based on serum creatinine values, as documentation of urine output is probably not sufficiently accurate. The creatinine measurements are part of routine clinical care. Therefore, absence of creatinine postoperative measurements are considered to be 'no suspicion of kidney injury'. KDIGO defines AKI as any of the following: Increase in serum creatinine by 0.3mg/dL or more within 48 hours or Increase in serum creatinine to 1.5 times baseline or more within the last 7 days or Urine output less than 0.5 mL/kg/h for 6 hours. Stage 1 is 1.5-9x baseline or >0.3 increase; Stage 2 is 2-2.9x baseline; Stage 3 is 3x baseline, or increase to > 4, or initiation of renal replacement therapy.
Time Frame: Within 7 days after surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants
  AKI stage II or greater | 1 | 0
  No stage II or greater - Confirmed by measurement | 11002 | 3157
  No postoperative creatinine measurement | 4621 | 1171

5. Secondary Outcome: Postoperative Rise in Creatinine Levels
Description: Absolute values for serum creatinine before and after surgery will be compared. When multiple postoperative creatinine measurements are made, the maximum difference is reported.
Time Frame: Within 7 days after surgery
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section). Patients with no routine postoperative creatinine measurements are excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 11003 | 3157
mg/dL | 0.00 [-0.10 to 0.13] | 0.00 [-0.09 to 0.14]

6. Secondary Outcome: Incidence of a MAP < 60 mmHg
Description: Incidence of a mean arterial pressure (MAP) < 60 mmHg during anesthesia for 1 minute or more.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 13779 | 3798

7. Secondary Outcome: Incidence of a MAP < 55 mmHg
Description: Incidence of a mean arterial pressure (MAP) < 55 mmHg during anesthesia for 1 minute or more.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 10991 | 3045

8. Secondary Outcome: Incidence of a MAP < 50 mmHg
Description: Incidence of a mean arterial pressure (MAP) < 50 mmHg during anesthesia for 1 minute or more.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 7781 | 2196

9. Secondary Outcome: Incidence of a MAP < 60 mmHg for > 10 Minutes
Description: Incidence of a mean arterial pressure (MAP) < 60 mmHg for a cumulative duration of all hypotensive episodes of more than 10 minutes during the anesthetic phase of the procedure.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 6989 | 1723

10. Secondary Outcome: Incidence of a MAP < 55 mmHg for > 10 Minutes
Description: Incidence of a mean arterial pressure (MAP) < 55 mmHg for a cumulative duration of all hypotensive episodes of more than 10 minutes during the anesthetic phase of the procedure.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 3181 | 759

11. Secondary Outcome: Incidence of a MAP < 50 mmHg for > 10 Minutes
Description: Incidence of a mean arterial pressure (MAP) < 50 mmHg for a cumulative duration of all hypotensive episodes of more than 10 minutes during the anesthetic phase of the procedure.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 1159 | 326

12. Secondary Outcome: Incidence of a MAP < 60 mmHg for > 20 Minutes
Description: Incidence of a mean arterial pressure (MAP) < 60 mmHg for a cumulative duration of all hypotensive episodes of more than 20 minutes during the anesthetic phase of the procedure.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 3632 | 792

13. Secondary Outcome: Incidence of a MAP < 55 mmHg for > 20 Minutes
Description: Incidence of a mean arterial pressure (MAP) < 55 mmHg for a cumulative duration of all hypotensive episodes of more than 20 minutes during the anesthetic phase of the procedure.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 1223 | 284

14. Secondary Outcome: Incidence of a MAP < 50 mmHg for > 20 Minutes
Description: Incidence of a mean arterial pressure (MAP) < 50 mmHg for a cumulative duration of all hypotensive episodes of more than 20 minutes during the anesthetic phase of the procedure.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 304 | 85

15. Secondary Outcome: Depth and Duration of Intraoperative Hypotension - Threshold MAP 75 mmHg
Description: Depth and duration of intraoperative hypotension will be modeled by calculating areas under the threshold for mean arterial pressures (MAPs). Thresholds will vary from 75 mmHg to 50 mmHg in 5 mmHg decrements. Together these variables represent the depth and duration of intraoperative hypotension. To optimize goodness of fit of these variables, the decremental steps may be increased to 10 mmHg and more restrictive lowest and highest thresholds may be chosen for the statistical analysis.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg*minute
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mmHg*minute | 485 [243 to 915] | 417 [206 to 764]

16. Secondary Outcome: Depth and Duration of Intraoperative Hypotension - Threshold MAP 70 mmHg
Description: as for outcome 15
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg*minute
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mmHg*minute | 273 [126 to 543] | 235 [109 to 451]

17. Secondary Outcome: Depth and Duration of Intraoperative Hypotension - Threshold MAP 65 mmHg
Description: as for outcome 15
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg*minute
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mmHg*minute | 96 [34 to 225] | 86 [30 to 193]

18. Secondary Outcome: Depth and Duration of Intraoperative Hypotension - Threshold MAP 60 mmHg
Description: as for outcome 15
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg*minute
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mmHg*minute | 57 [21 to 131] | 52 [20 to 117]

19. Secondary Outcome: Depth and Duration of Intraoperative Hypotension - Threshold MAP 55 mmHg
Description: as for outcome 15
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg*minute
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mmHg*minute | 23 [5 to 59] | 23 [5 to 62]

20. Secondary Outcome: Depth and Duration of Intraoperative Hypotension - Threshold MAP 50 mmHg
Description: as for outcome 15
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg*minute
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mmHg*minute | 19 [7 to 43] | 19 [8 to 47]

21. Secondary Outcome: Estimated Intraoperative Blood Loss
Description: The estimated blood loss in mL during the surgical procedure
Time Frame: During the surgical procedure: an expected average of 2 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mL | 100 [25 to 250] | 75 [20 to 200]

22. Secondary Outcome: Time to Discharge Readiness at the Postanesthesia Care Unit (PACU)
Description: The time from arriving at the postanesthesia care unit (PACU) until the time the patient is considered ready for discharge (in minutes).
Time Frame: A specific time frame on the day of surgery: from the start of admission to the PACU to discharge from the PACU, an expected average of 4 hours
Population: Only patients with a postoperative stay at the postanesthesia care unit (PACU). Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section).
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 13082 | 3580
minutes | 67 [46 to 101] | 60 [42 to 89.25]

23. Secondary Outcome: Intravenous Anesthetic Drug Use During Intraoperative Hypotension: MAP < 65 mmHg
Description: Average concentrations of propofol infusion rates during MAP < 65 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 65 mmHg and a continuous administration of one of the following anesthetics: propofol, sevoflurane, isoflurane, desflurane. On occasion, the anesthesiologist may switch between anesthetic drugs. The numbers analyzed in one or more rows thus does not match the overall number analyzed.
Measure: Median (Inter-Quartile Range); unit: mcg/kg/min (propofol)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 14333 | 3926
mcg/kg/min (propofol) | 60.10 [35 to 100] | 48.59 [28.55 to 83.88]

24. Secondary Outcome: Intravenous Anesthetic Drug Use During Intraoperative Hypotension: MAP < 60 mmHg
Description: Average concentrations of propofol infusion rates during MAP < 60 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 60 mmHg and either a continuous administration of one of the following anesthetics: propofol, sevoflurane, isoflurane, desflurane. On occasion, the anesthesiologist may switch between anesthetic drugs. The numbers analyzed in one or more rows thus does not match the overall number analyzed.
Measure: Median (Inter-Quartile Range); unit: mcg/kg/min (propofol)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 11621 | 3145
mcg/kg/min (propofol) | 61.07 [37.39 to 100.00] | 50.00 [27.65 to 81.50]

25. Secondary Outcome: Intravenous Anesthetic Drug Use During Intraoperative Hypotension: MAP < 55 mmHg
Description: Average concentrations of propofol infusion rates during MAP < 55 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 55 mmHg and either a continuous administration of one of the following anesthetics: propofol, sevoflurane, isoflurane, desflurane. On occasion, the anesthesiologist may switch between anesthetic drugs. The numbers analyzed in one or more rows thus does not match the overall number analyzed.
Measure: Median (Inter-Quartile Range); unit: mcg/kg/min (propofol)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 8254 | 2196
mcg/kg/min (propofol) | 63.95 [37.50 to 100.00] | 50.00 [29.12 to 83.33]

26. Secondary Outcome: Intravenous Anesthetic Drug Use During Intraoperative Hypotension: MAP < 50 mmHg
Description: Average concentrations of propofol infusion rates during MAP < 50 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 50 mmHg and a continuous administration of one of the following anesthetics: propofol, sevoflurane, isoflurane, desflurane. On occasion, the anesthesiologist may switch between anesthetic drugs. The numbers analyzed in one or more rows thus does not match the overall number analyzed.
Measure: Median (Inter-Quartile Range); unit: mcg/kg/min (propofol)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 5135 | 1413
mcg/kg/min (propofol) | 65.00 [40.00 to 100.00] | 50.00 [30.00 to 82.71]

27. Secondary Outcome: Average Use of Cardiovascular Drugs: Ephedrine
Description: Cardiovascular drugs as defined under interventions. Average use for each drug will be calculated. Cardiovascular drugs that were given in <1% of cases are not reported, as the average dosages would be meaningless.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section). In addition, only patients that actually received any ephedrine are analyzed.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 9310 | 2718
mg | 20 [10 to 25] | 15 [10 to 25]

28. Secondary Outcome: Average Use of Cardiovascular Drugs: Phenylephrine
Description: Cardiovascular drugs as defined under interventions. Average use for each drug will be calculated. Cardiovascular drugs that were given in <1% of cases are not reported, as the average dosage would be meaningless.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section). In addition, only patients that actually received any phenylephrine are analyzed.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 12211 | 3685
mg | 0.90 [0.30 to 3.69] | 1.30 [0.40 to 5.03]

29. Secondary Outcome: Average Use of Cardiovascular Drugs: Glycopyrrolate
Description: as for outcome 28
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section). In addition, only patients that actually received any glycopyrrolate are analyzed.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 11093 | 1257
mg | 0.40 [0.40 to 0.60] | 0.40 [0.20 to 0.40]

30. Secondary Outcome: Average Use of Cardiovascular Drugs: Epinephrine
Description: as for outcome 28
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section). In addition, only patients that actually received any epinephrine are analyzed.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 1215 | 409
mg | 1.00 [0.50 to 2.00] | 0.70 [0.50 to 2.00]

31. Secondary Outcome: Average Use of Cardiovascular Drugs: Norepinephrine
Description: as for outcome 28
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: Per study protocol only patients with any MAP < 65 mmHg will be included in the primary analysis (See also 'Participant Flow' section). In addition, only patients that actually received any norepinephrine are analyzed.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 762 | 233
mg | 0.62 [0.27 to 1.35] | 0.70 [0.33 to 1.56]

32. Secondary Outcome: Timing of Cardiovascular Drugs for MAP < 65 mmHg
Description: Cardiovascular drugs as defined under interventions. Time of first administration of cardiovascular drug relative to the time at which the mean arterial pressure (MAP) drops below 60 mmHg. Per patient the average time to first administration of all hypotensive episodes was calculated. That average time is used as the outcome variable. A negative value indicates that administration occurred before the drop in MAP.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 65 mmHg and an administration event of a cardiovascular drugs within 5 minutes before the start of the hypotensive episode (the first value below 65 mmHg) and 15 minutes after the start of the episode.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 13932 | 3975
minutes | 2 [0.4 to 4] | 1.14 [0 to 3]

33. Secondary Outcome: Timing of Cardiovascular Drugs for MAP < 60 mmHg
Description: as for outcome 32
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 60 mmHg and an administration event of a cardiovascular drugs within 5 minutes before the start of the hypotensive episode (the first value below 60 mmHg) and 15 minutes after the start of the episode.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 12292 | 3458
minutes | 0.8 [-0.370 to 2.5] | 1.5 [0 to 3.5]

34. Secondary Outcome: Timing of Cardiovascular Drugs for MAP < 55 mmHg
Description: Cardiovascular drugs as defined under interventions. Time of first administration of cardiovascular drug relative to the time at which the mean arterial pressure (MAP) drops below 55 mmHg. Per patient the average time to first administration of all hypotensive episodes was calculated. That average time is used as the outcome variable. A negative value indicates that administration occurred before the drop in MAP.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 55 mmHg and an administration event of a cardiovascular drugs within 5 minutes before the start of the hypotensive episode (the first value below 55 mmHg) and 15 minutes after the start of the episode.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 9706 | 2752
minutes | 1 [-0.333 to 3] | 0.5 [-0.75 to 2.33]

35. Secondary Outcome: Timing of Cardiovascular Drugs for MAP < 50 mmHg
Description: Cardiovascular drugs as defined under interventions. Time of first administration of cardiovascular drug relative to the time at which the mean arterial pressure (MAP) drops below 50 mmHg. Per patient the average time to first administration of all hypotensive episodes was calculated. That average time is used as the outcome variable. A negative value indicates that administration occurred before the drop in MAP.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: All patients with any MAP < 50 mmHg and an administration event of a cardiovascular drugs within 5 minutes before the start of the hypotensive episode (the first value below 50 mmHg) and 15 minutes after the start of the episode.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 6789 | 1989
minutes | 1 [-0.833 to 3] | 0 [-1 to 2.17]

36. Secondary Outcome: Intraoperative Administration of Intravenous Fluids
Description: Total amount (mL) of intravenous fluids (as defined under interventions) administered during the surgical procedure.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
mL | 1500.00 [1000.00 to 2300.00] | 1400.00 [1000.00 to 2000.00]

37. Post Hoc Outcome: Postoperative Acute Kidney Injury
Description: as for outcome 1
Time Frame: Within 7 days after surgery
Population: Post-Hoc analysis: all patients, not only those with any MAP < 65 mmHg.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 17463 | 4972
Participants
  AKI stage I or greater | 1477 | 435
  No AKI - Confirmed by measurement | 10690 | 3166
  No postoperative creatinine measurement | 5296 | 1371

38. Post Hoc Outcome: Usage Frequency of Cardiovascular Drugs: Ephedrine
Description: Cardiovascular drugs as defined under interventions. Frequency of patients receiving the drug. Cardiovascular drugs that were given in <1% of cases are not reported.
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 9310 | 2718

39. Post Hoc Outcome: Usage Frequency of Cardiovascular Drugs: Phenylephrine
Description: as for outcome 38
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 12211 | 3685

40. Post Hoc Outcome: Usage Frequency of Cardiovascular Drugs: Glycopyrrolate
Description: as for outcome 38
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 11093 | 1257

41. Post Hoc Outcome: Usage Frequency of Cardiovascular Drugs: Ephinephrine
Description: as for outcome 38
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 1215 | 409

42. Post Hoc Outcome: Usage Frequency of Cardiovascular Drugs: Norepinephrine
Description: as for outcome 38
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 15624 | 4328
Participants | 762 | 233

43. Secondary Outcome: Inhaled Anesthetic Drug Use During Intraoperative Hypotension: MAP < 65 mmHg
Description: Average concentrations of inhalational anesthesia during MAP < 65 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: EndTidal% (other)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 14333 | 3926
EndTidal% (other)
  Sevoflurane (EndTidal %): number analyzed (Participants) | 4589 | 1258
  Sevoflurane (EndTidal %) | 1.35 [1.03 to 1.6] | 1.27 [0.98 to 1.55]
  Isoflurane (EndTidal %): number analyzed (Participants) | 9325 | 2522
  Isoflurane (EndTidal %) | 0.68 [0.56 to 0.80] | 0.68 [0.56 to 0.80]
  Desflurane (EndTidal %): number analyzed (Participants) | 63 | 2
  Desflurane (EndTidal %) | 4.10 [3.31 to 4.64] | 2.31 [1.15 to 3.46]

44. Secondary Outcome: Inhaled Anesthetic Drug Use During Intraoperative Hypotension: MAP < 60 mmHg
Description: Average concentrations of inhalational anesthesia during MAP < 60 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: EndTidal% (other)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 11621 | 3145
EndTidal% (other)
  Sevoflurane (EndTidal %): number analyzed (Participants) | 3656 | 997
  Sevoflurane (EndTidal %) | 1.35 [1.02 to 1.62] | 1.25 [0.95 to 1.57]
  Isoflurane (EndTidal %): number analyzed (Participants) | 7400 | 1949
  Isoflurane (EndTidal %) | 0.68 [0.55 to 0.80] | 0.67 [0.55 to 0.80]
  Desflurane (EndTidal %): number analyzed (Participants) | 50 | 2
  Desflurane (EndTidal %) | 4.36 [3.40 to 4.80] | 2.33 [1.116 to 3.49]

45. Secondary Outcome: Inhaled Anesthetic Drug Use During Intraoperative Hypotension: MAP < 55 mmHg
Description: Average concentrations of inhalational anesthesia during MAP < 55 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: EndTidal% (other)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 8254 | 2196
EndTidal% (other)
  Sevoflurane (EndTidal %): number analyzed (Participants) | 2551 | 706
  Sevoflurane (EndTidal %) | 1.34 [1.00 to 1.62] | 1.25 [0.94 to 1.55]
  Isoflurane (EndTidal %): number analyzed (Participants) | 5099 | 1294
  Isoflurane (EndTidal %) | 0.68 [0.52 to 0.82] | 0.67 [0.52 to 0.80]
  Desflurane (EndTidal %): number analyzed (Participants) | 31 | 1
  Desflurane (EndTidal %) | 4.60 [3.49 to 4.88] | 4.65 [4.65 to 4.65]

46. Secondary Outcome: Inhaled Anesthetic Drug Use During Intraoperative Hypotension: MAP < 50 mmHg
Description: Average concentrations of inhalational anesthesia during MAP < 50 mmHg episodes
Time Frame: During the anesthetic phase of the surgical procedure: an expected average of 2.5 hours
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: EndTidal% (other)
Arm/Group | Usual Care Group | Hypotension Decision Support
Number analyzed (Participants) | 5135 | 1413
EndTidal% (other)
  Sevoflurane (EndTidal %): number analyzed (Participants) | 902 | 400
  Sevoflurane (EndTidal %) | 1.32 [1.00 to 1.65] | 1.23 [0.89 to 1.57]
  Isoflurane (EndTidal %): number analyzed (Participants) | 3067 | 799
  Isoflurane (EndTidal %) | 0.65 [0.50 to 0.82] | 0.65 [0.50 to 0.80]
  Desflurane (EndTidal %): number analyzed (Participants) | 16 | 1
  Desflurane (EndTidal %) | 4.28 [3.61 to 4.78] | 4.70 [4.70 to 4.70]

ADVERSE EVENTS:
Time Frame: We analyzed adverse events in this patient population during their intraoperative course (adverse events sourced from our adverse event reporting system; from entry into OR to exit from OR), and during their hospitalization (source for mortality data; from hospital admission to hospital discharge).
Description: We utilized our perioperative information management system to determine the number of adverse events that occurred associated with the patients' intraoperative course. We used our hospital registration system to determine all cause mortality for this patient population.
Arm/Group | Usual Care Group | Hypotension Decision Support
All-Cause Mortality (participants affected / at risk) | 534/17463 | 158/4972
Serious Adverse Events (participants affected / at risk) | 1811/17463 | 541/4972
Other Adverse Events (participants affected / at risk) | 0/17463 | 0/4972
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care Group (N=17463) | Hypotension Decision Support (N=4972)
Acute Kidney Injury Stage I or greater (Renal and urinary disorders) | 1477 | 435 — KDIGO (Kidney Disease: Improving Global Outcomes) Stage I or greater within the first seven postoperative days of surgery. Only based on creatinine measurements as part of routine clinical care, not urine output (inadequate documentation).
Mortality (Investigations) | 534 | 158

LIMITATIONS AND CAVEATS:
1. Due to development issues the UMC Utrecht could not participate: myocardial injury was dropped as primary outcome, as well as some secondary outcomes.
2. Technical issues at the VUMC resulted in absent IOH notifications (see 'Participant Flow').

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT02726620/Prot_SAP_000.pdf